CLINICAL TRIAL: NCT00469963
Title: Clinical Trial of Sir Spheres® in Patients With Primary Hepatocellular Carcinoma
Brief Title: Internal Radiation Therapy in Treating Patients With Primary Liver Cancer That Cannot Be Removed by Surgery
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: slow accrual
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Steven Meranze, MD, Vice-Chair, Department of Radiology and Radiological Science; Professor of Radiology and Surgery; Interventional Radiologist, Vanderbilt-Ingram Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VICC GI 0364; VU-VICC-GI-0364
Record Dates: First submitted 2007-05-03; First posted 2007-05-07 (Estimated); Last update posted 2012-09-03 (Estimated); Status verified 2012-08

CONDITIONS: Liver Cancer
Keywords: adult primary hepatocellular carcinoma; localized unresectable adult primary liver cancer; recurrent adult primary liver cancer; advanced adult primary liver cancer
MeSH Terms: conditions — Liver Neoplasms; Carcinoma, Hepatocellular | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- SIR-SPHERES (Experimental)
  Interventions: Procedure: quality-of-life assessment; Radiation: yttrium Y 90 resin microspheres

INTERVENTIONS:
Procedure: quality-of-life assessment — quality-of-life assessment
Radiation: yttrium Y 90 resin microspheres — radiation therapy
  Other Names: radiation therapy

SUMMARY:
RATIONALE: Specialized internal radiation therapy that delivers a high dose of radiation directly to the tumor may kill more tumor cells and cause less damage to normal tissue.

PURPOSE: This clinical trial is studying how well internal radiation therapy works in treating patients with primary liver cancer that cannot be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine tumor response to selective internal radiation therapy comprising yttrium Y 90 resin microspheres (Sir-Spheres®) in patients with unresectable primary hepatocellular carcinoma.

Secondary

* Determine the toxicity of this regimen in these patients.
* Determine the health-related quality of life of patients receiving this regimen.
* Determine the survival of patients receiving this regimen.

OUTLINE: Patients undergo selective internal radiation therapy comprising yttrium Y 90 resin microspheres (Sir-Spheres®) via catheter directly into the hepatic artery on day 1.

Health-related quality of life is assessed prior to initial treatment and then periodically thereafter.

After completion of study treatment, patients are followed periodically for 12-24 months.

PROJECTED ACCRUAL: A total of 35 patients will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of hepatocellular carcinoma

  * Not amenable to surgical resection or immediate liver transplantation

    * Destaging of tumor prior to surgical resection or transplantation allowed
* Measurable disease, defined as ≥ 1 lesion that can be accurately measured in ≥ 1 dimension (longest diameter to be recorded) ≥ 10 mm by contrasted CT scan

  * No equivocal, nonmeasurable, or nonevaluable liver cancer
* No more than 75% replacement of normal liver by tumor
* Cancer of the Liver Italian Program (CLIP) stage 1-3 disease
* No extra-hepatic metastases as determined by CT scan or MRI

Exclusion Criteria:

* Life expectancy ≥ 3 months
* Karnofsky performance status 50-100%
* Creatinine ≤ 1.5 mg/dL
* Bilirubin ≤ 2.0 mg/dL
* Albumin ≥ 3 g/dL
* Granulocyte count ≥ 1,500/mm³
* Platelet count ≥ 65,000/mm³
* INR ≤ 1.4
* Hemoglobin > 9 g/dL
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 3 months after completion of study treatment
* No nonmalignant disease that would render the patient ineligible for treatment according to this protocol
* No hepatic arterial anatomy that would prevent the administration of study drug into the liver
* Less than 20% arteriovenous lung shunting on a technetium 99m-labeled macroaggregated albumin nuclear scan
* No other malignancy within the past 5 years except for cured basal cell carcinoma of the skin or cured carcinoma in situ of the uterine cervix

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* More than 90 days since prior surgery, chemotherapy, or locally ablative technique for the liver cancer
* More than 4 weeks since prior and no other concurrent investigational drug or agent/procedure (i.e., participation in another trial)
* No prior radiotherapy to the upper abdomen that included the liver in the treatment field
* No capecitabine within 8 weeks before or after study treatment
* No other anticancer treatment (except surgical resection) for liver cancer during and for 3 months after completion of study treatment

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2003-12; Primary Completion 2006-10 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Tumor response | up to 12 months
  All uni-dimensional measurable lesions (longest diameter >20mm with conventional techniques and >10mm with spiral CT scans) up to a maximum of five lesions per organ with a maximum of 10 lesions in total are used to determine response.

SECONDARY OUTCOMES:
Toxicity | up to 3 months
Health-related quality of life | prior to initial treatment.
  The assessment will include a Karnofsky score the patient-completed SF-36 questionnaire. This information will be assessed at each quarterly evaluation, as well as any unscheduled clinical appointments. Karnofsky functional performance36 will be assessed by a clinician. This widely-used scale ranges from 0 to 100 and derives three broad categories of functional performance (able: 80-100; unable: 50-70; and disabled: 0-40).
  Patient report of HRQOL will be determined via the Medical Outcome Study 36-item short form (SF-36)37, which includes eight individual scales, physical and mental component summary scores, and is normed to both healthy and clinical populations.
Survival | trial entry to death

CONTACTS AND LOCATIONS:
Overall Officials: Steven G. Meranze, MD, Principal Investigator — Vanderbilt-Ingram Cancer Center
Locations (1):
- Vanderbilt-Ingram Cancer Center, Nashville, Tennessee, United States